CLINICAL TRIAL: NCT05256888
Title: Time-Restricted Eating to Address Persistent Cancer-Related Fatigue: The Fatigue REDuction After Cancer (FREDA) Trial
Brief Title: Time-Restricted Eating to Address Persistent Cancer-Related Fatigue
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Amber Kleckner, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00099067; UL1TR003098 (NIH)
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Neoplasms; Therapy; Fatigue; Diet Therapy; Time; Survivorship; Fasting, Intermittent
MeSH Terms: conditions — Neoplasms; Fatigue; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating (Experimental): Participants will self-select a 10-hour window in which to consume all food and beverages (with the exception of black coffee and unsweetened tea in the mornings; water is okay at all times). Participants will also receive weekly tips to encourage a healthy lifestyle in cancer survivorship.
  Interventions: Behavioral: Time-restricted eating; Behavioral: Healthy lifestyle education
- Control (Other): Participants will receive weekly tips to encourage healthy lifestyle behaviors in cancer survivorship.
  Interventions: Behavioral: Healthy lifestyle education

INTERVENTIONS:
Behavioral: Time-restricted eating — 12 weeks of time-restricted eating (10-hour window)
  Arms: Time-restricted eating
Behavioral: Healthy lifestyle education — Weekly tips on healthy lifestyle behaviors (e.g., diet, exercise, sleep) for 12 weeks

SUMMARY:
This study will assess the feasibility of delivering a 12-week time-restricted eating intervention as well as the intervention's preliminary efficacy on persistent cancer-related fatigue among cancer survivors compared to a general health education control. Participants will be randomized 1:1 to one of two arms: time-restricted eating or control. Those in the intervention arm will self-select a 10-hour eating window in which to consume all food and beverages (water is allowed any time, black coffee and unsweetened tea are allowed in the morning). Both groups will receive weekly educational tips on healthy lifestyle behaviors in cancer survivorship. This study will also explore relationships between fatigue, circadian rhythm, and glucose metabolism.

The hypothesis is that recruitment will be feasible, and participants will adhere to time-restricted eating and complete study activities over the course of the 12 weeks. The second hypothesis is that time-restricted eating will lead to less fatigue at 12 weeks compared to the control, accounting for baseline fatigue levels.

ELIGIBILITY:
Inclusion Criteria:

* Have completed adjuvant chemotherapy, surgery, and/or radiation for cancer, including chemotherapy for hematologic neoplasms, at least 2 months and not more than 2 years prior to enrolling,
* Have a baseline level of fatigue, as determined by reporting a score of 4 or higher for the question, "In the last week, how bad was your worst fatigue on a scale from 0-10?"
* Be able to speak and/or read and write in English,
* Be at least 18 years old,
* Own a smartphone,
* Be willing and able to adhere to study procedures, including use of a smartphone app, and
* Be able to provide informed consent.

Exclusion Criteria:

* Already eat all their food within a window that is 10 h or shorter most (6/7) days of the week,
* Be underweight, as defined as a body mass index ≤18.5 kg/m2,
* Have surgery planned during the study duration,
* Have any contraindications to the proposed nutrition intervention as identified by their medical provider, their designee, or the study team (e.g., type 1 diabetes, risk for hypoglycemia, medication requirements, pregnancy, breastfeeding, recent history of an eating disorder),
* Be taking insulin, or
* Be on enteral or parenteral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2026-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Kleckner AS, Clingan CL, Youngblood SM, Kleckner IR, Quick L, Elrod RD, Zhu S, Manoogian ENC, Panda S, Badros AZ, Emadi A. Time-restricted eating to address persistent cancer-related fatigue among cancer survivors: a randomized controlled trial. Support Care Cancer. 2025 Apr 5;33(4):353. doi: 10.1007/s00520-025-09394-w. PMID 40186671

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants must have completed baseline assessments, including the FACIT-F questionnaire, in order to be randomized. There were 20 people who consented to the study but did not complete baseline assessments and therefore were not randomized to an arm.
Period: Overall Study
Arm/Group | Time-restricted Eating | Control
Started | 15 | 15
Completed | 14 | 11
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Time-restricted Eating | Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (12.7) | 53.7 (16.8) | 54.1 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 13 | 15 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 6 | 16
  White | 5 | 8 | 13
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility, as Assessed by the Percentage of Participants Who Enrolled Completed the Study
Description: To assess feasibility, the percentage of participants who provide evaluable data regarding their eating window at baseline and 12 weeks will be assessed.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants
Arm/Group | All Participants
Number analyzed (Participants) | 50
Participants | 25

2. Primary Outcome: Fatigue, as Assessed Using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Questionnaire
Description: FACIT-F fatigue subscale scores will be compared for those in the time-restricted eating group vs. the control group at week 12, controlling for baseline levels. This questionnaire is 13-items long. The scale is from 0-52, and a higher score indicates less fatigue.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Time-restricted Eating | Control
Number analyzed (Participants) | 11 | 14
score on a scale | 38.7 (9.2) | 37.2 (9.1)
Statistical Analysis 1: Comparison: Time-restricted Eating vs Control; In a linear model to assess group effects on fatigue at 12 weeks, adjusting for baseline levels of fatigue: Effect of group = -1.77±1.08, p=0.11, favoring the TRE group; Test type: Superiority; p = 0.11, Regression, Linear; Slope = -1.77, Standard Error of Mean 1.08

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Time-restricted Eating | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Time-restricted Eating (N=15) | Control (N=15)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Time-restricted Eating (N=15) | Control (N=15)
Nausea and diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT05256888/Prot_SAP_ICF_000.pdf